CLINICAL TRIAL: NCT07323459
Title: Effectiveness of an Individual Midwife-Led Psychoeducational Intervention in Reducing Pregnancy-Related Anxiety in Pregnant Women
Brief Title: A Midwife-Led Psychoeducational Intervention to Reduce Pregnancy-Related Anxiety in Low-Risk Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KB/367/2025
Record Dates: First submitted 2025-12-08; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy-Related Anxiety (PrA); Fear of Childbirth
Keywords: prenatal care; pregnancy-related anxiety; maternal mental health; anxiety; pregnancy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant women with high PrA levels receiving midwife-led individual psychoeducational intervention (Experimental)
  Interventions: Other: A Midwife-Led Psychoeducational Intervention to Reduce Pregnancy-Related Anxiety in Low-Risk Pregnant Women
- Standard prenatal care without additional psychoeducational intervention (No Intervention)

INTERVENTIONS:
Other: A Midwife-Led Psychoeducational Intervention to Reduce Pregnancy-Related Anxiety in Low-Risk Pregnant Women — Individual program by midwife in 2nd/3rd trimester: 4-6 sessions (~60min), every 1-2 weeks.
  Session 1: PRAQ-R2 assessment, identifying fears, building trust. Session 2: Labor stages education, myth verification, visual aids. For multiparous: previous birth discussion.
  Session 3: Pain management - breathing, relaxation, massage, hydrotherapy, epidural, nitrous oxide. Practical exercises.
  Session 4: Birth plan development, assertive communication training, role-playing.
  Session 5: Mindfulness, cognitive restructuring, affirmations, visualization, final PRAQ-R2.
  Session 6 (optional): Techniques review, birth plan finalization, Q&A, contact plan.
  Materials: brochures, diagrams, videos, templates, audio instructions. Flexible, individualized.
  Arms: Pregnant women with high PrA levels receiving midwife-led individual psychoeducational intervention

SUMMARY:
The goal of this clinical trial is to evaluate whether an individualized psychoeducational intervention led by an experienced midwife can reduce pregnancy-related anxiety (PrA) in pregnant women during the second and third trimesters. The main questions it aims to answer are:

* Can individualized midwife-led psychoeducation significantly reduce pregnancy-related anxiety levels as measured by the PRAQ-R2 questionnaire?
* Does this intervention improve women's sense of control, competence, and readiness for childbirth?
* Can the intervention reduce preferences for cesarean section without medical indication among low-risk pregnant women?

Participants will:

* Attend 4-6 individual sessions (approximately 60 minutes each) with a midwife, scheduled every 1-2 weeks
* Complete the Pregnancy-Related Anxiety Questionnaire (PRAQ-R2) at the beginning and end of the intervention to measure anxiety levels
* Receive evidence-based education about the physiological process of childbirth, pain management methods (both pharmacological and non-pharmacological), and medical procedures
* Learn and practice stress-reduction techniques including breathing exercises, relaxation methods, and mindfulness
* Develop an individualized birth plan and practice communication skills for effective interaction with medical personnel
* Work on cognitive strategies to address negative thoughts and build positive affirmations about childbirth

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the second or third trimester of pregnancy
* Elevated level of pregnancy-related anxiety (PrA)
* Low obstetric risk pregnant women (no significant medical contraindications to vaginal delivery)
* Consent to participate in individual psychoeducational sessions
* Ability to communicate in Polish at a level sufficient to understand the materials and participate in the sessions

Exclusion Criteria:

* Pregnant women with severe mental disorders requiring urgent psychiatric intervention
* Women with serious obstetric complications in the current pregnancy requiring intensive medical monitoring (e.g., severe hypertension, imminent preterm delivery requiring hospitalization)
* Patients already undergoing intensive psychotherapy or pharmacotherapy for anxiety
* Lack of consent to participate or inability to attend sessions (e.g., due to logistical reasons)
* Pregnant women whose pregnancy-related anxiety is not the primary concern, with other dominant anxiety disorders (e.g., GAD unrelated to pregnancy) or other priority health needs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Pregnancy-Related Anxiety Level | Baseline (Session 1, before intervention start) and post-intervention (after completing 4-6 sessions, approximately 8-12 weeks from baseline)
  Measure: Change in Pregnancy-Related Anxiety Questionnaire-Revised 2 (PRAQ-R2) total score from baseline to post-intervention.
  Description: The PRAQ-R2 is a validated 10-item questionnaire assessing pregnancy-specific anxiety, using a 5-point Likert scale. Total scores range from 10 to 50, with higher scores indicating higher levels of pregnancy-related anxiety (worse outcome). The Polish validated version of the questionnaire will be used. A decrease in score reflects a reduction in anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Obstetric and Gynaecological Nursing, Faculty of Health Sciences with the Institute of Maritime and Tropical Medicine, Medical University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect participant confidentiality and due to data protection regulations. Results will be published in aggregated form.